CLINICAL TRIAL: NCT04382846
Title: Nitazoxanide in Treatment of COVID-19
Brief Title: Novel Regimens in COVID-19 Treatment
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tanta covid treatment
Record Dates: First submitted 2020-05-07; First posted 2020-05-11 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: COVID; Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — nitazoxanide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide (Experimental): Nitazoxanide with standard protocol of treatment
  Interventions: Drug: Nitazoxanide
- Control group (No Intervention): Standard protocol alone

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide
  Other Names: Parazoxanide, Nanazoxid
  Arms: Nitazoxanide

SUMMARY:
Nitazoxanide has been shown to have a clinical efficacy against severe acute respiratory syndrome coronavirus 2; ivermectin has also demonstrated a remarkable experimental efficacy with a potential to be used for Coronavirus disease 2019.

DETAILED DESCRIPTION:
Nitazoxanide has been shown to have a clinical efficacy against severe acute respiratory syndrome coronavirus; ivermectin has also demonstrated a remarkable experimental efficacy with a potential to be used for Coronavirus disease 2019. Some studies demonstrated the efficacy of combined regimen of nitazoxanide and azithromycin or ivermectin and chloroquine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COVID-19 infection

Exclusion Criteria:

* Allergy or contraindication to the drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with virological cure | 6 months
  the number of patients with virological cure

CONTACTS AND LOCATIONS:
Overall Officials: sherief Abd-Elsalam, Ass. Prof., Principal Investigator — ass. Prof. Tropical Medicine
Locations (2):
- Egypt (2):
  - Tanta University, Assiut University, Tanta
  - Sherief Abd-Elsalam, Tanta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelleni MT. Nitazoxanide/azithromycin combination for COVID-19: A suggested new protocol for early management. Pharmacol Res. 2020 Jul;157:104874. doi: 10.1016/j.phrs.2020.104874. Epub 2020 Apr 30. PMID 32360581
- [Background] Choudhary R, Sharma AK. Potential use of hydroxychloroquine, ivermectin and azithromycin drugs in fighting COVID-19: trends, scope and relevance. New Microbes New Infect. 2020 Apr 22;35:100684. doi: 10.1016/j.nmni.2020.100684. eCollection 2020 May. PMID 32322397